CLINICAL TRIAL: NCT02108613
Title: Living Well on Androgen Deprivation Therapy: A Comprehensive Approach to Prostate Cancer Survivorship
Brief Title: Living Well on Androgen Deprivation Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: It was deemed not enough funding and the initial funding returned and study withdrawn (never opened and no recruitment happened.
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: The Prostate Centre - Vancouver Island and the Gulf Islands (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 084902
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2014-04

CONDITIONS: Prostate Cancer
Keywords: Androgen deprivation therapy; Supportive care; Quality of life
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): The intervention arm will receive sexual health counselling, exercise sessions, nutrition education, and will be assigned a peer support volunteer.
  Interventions: Behavioral: Exercise Sessions; Behavioral: Nutrition Education; Behavioral: Peer Support Volunteer
- Control (No Intervention): The control group will receive sexual health counseling.

INTERVENTIONS:
Behavioral: Exercise Sessions — 8 weeks of weekly exercise classes taught by a certified exercise physiologist.
  Arms: Intervention
Behavioral: Nutrition Education — Four monthly education sessions on nutrition topics. Presentations and materials are were created by a BCCA dietitian.
  Arms: Intervention
Behavioral: Peer Support Volunteer — Participants will be assigned a peer support volunteer who will preform adherence calls to discuss goals and motivations about improving exercise and healthy eating.
  Arms: Intervention

SUMMARY:
Approximately half of men treated for prostate cancer will be offered hormone deprivation therapy during their cancer experience. The secondary effects of this treatment can result in osteoporosis, cardiovascular disease, stroke, diabetes, and diminished sexual health. To promote healthy lifestyle choices for couples and maintain their intimacy and emotional health we propose the Living Well, an innovative program that combines nutrition, physical activity, and sexual health initiatives in one integrated service. This project will be piloted at the Vancouver Island Centre with an expected 100 patients over 1 year. Over a six month period both the experimental and control groups will have access to a workbook (designed for men with prostate cancer and on hormone deprivation therapy) and sexual health counseling. The experimental group will also have access to an exercise and a nutritional program and support by volunteers to keep motivated. Assessment will look at quality of life, physical factors, and biomarkers associated with secondary disease.

DETAILED DESCRIPTION:
1. Purpose:

   The overarching goal of the Living Well project is to maintain or improve quality of life for people with prostate cancer on androgen deprivation therapy (ADT) and their partners by providing the couples with the tools to promote confidence and motivation to remain both physically and psychosocially healthy and intimate. The primary objective is to determine the effect of our comprehensive community-based survivorship program on psychosocial health of people with PCa on ADT and their partners. Secondarily we intend to explore the impact of the program on biomarkers associated with the metabolic syndrome often observed in men on ADT, the program's operational and perceived (by patients and partners) impact of the program.
2. Hypothesis:

   1. The intervention group will show a larger magnitude of improvement on measures of QOL, fatigue, and intimacy, ultimately leading to increased benefit when compared to the control group.
   2. We believe through the engagement of peer volunteers that compliance and adherence to positive lifestyle changes will be higher on the intervention group when compared to the control group.
3. Justification:

   ADT has offered people with prostate cancer (PCa) improved curative outcomes when combined with local radiation therapy and has been fundamental in controlling disease for those with a biochemical recurrence or metastatic disease. Due to its effectiveness, ADT is offered to up to 50% of people with PCa.

   ADT reduces the occurrence of metastases by lowering testosterone levels. Unfortunately, decreased testosterone can lead to hot flashes, diminished libido, erectile dysfunction, depression, diminished muscle strength, reduced bone mineral density, increased fat mass, and increased cholesterol levels. This conglomerate of secondary effects can lead to osteoporosis, cardiovascular disease, stroke, and diabetes. Poor lifestyle habits can further aggravate these secondary effects of ADT therapy. Being overweight may increase the risk of mortality from PCa. However, the increase in vascular disease and diabetes seems to be more strongly correlated with death than the cancer itself. Those with pre-existing cardiac problems and receiving ADT, have a 75% chance of dying from cardiovascular disease rather than PCa.

   There is growing evidence that healthy lifestyle practices that include a healthy diet and regular physical activity can improve the overall prognosis of PCa patients and diminish the negative effects of ADT. Many cancer survivors are motivated to seek information about food choices and physical activity to improve their response to treatment and quality of life. Recent research has shown that a preemptive educational program built around a book, the "Androgen Deprivation Therapy: An Essential Guide for Prostate Cancer Patients and Their Loved Ones", or the "Workbook" for short, which addresses all issues of life style management, can be effective in helping patients and their families in overcoming the challenges of ADT.

   The Workbook was created by a national team of PCa experts (the ADT Working Group) and is endorsed by the Canadian Urological Association. The Workbook addresses the well-established, physical and emotional adverse effects of ADT. Although not all ADT side effects directly reduce a patient's survival, they may greatly impact a patient and his partner's QoL. Important aspects explored in the Workbook include the psychosocial effects of ADT, exercise needs, and the nutritional recommendations for men on ADT. Previous research indicates that the effectiveness of the Workbook is enhanced when distributed to patients prior to the start of ADT, before side effects manifest. The Workbook's effectiveness is also enhanced when combined with motivational sessions led by trained educators.

   Given that people with PCa on ADT and their partners generally struggle with aspects of their sexual health, nutrition, and physical activity concurrently, we propose for the first time to test a comprehensive PCa survivorship approach, the Living Well program, which addresses concerns related to all three components. This is a community-based program designed for PCa patients prior to starting on ADT and will also be extended to their partners. The program will make extensive use of the ADT Workbook and will be primarily delivered using existing resources.
4. Objectives:

   The primary outcomes are:
   * Quality of Life
   * Fatigue

   Secondary outcome is

   - Intimacy

   We will also explore:
   * Effects on biomarkers associated with the metabolic syndrome secondary to ADT *
   * Effects on erectile dysfunction, PSA and testosterone levels*
   * The perceptions of patients and partners about the impact of the program on their psychosocial health
   * Operational impact

   Note: *Patient's health records will be checked to obtain annual blood measures of cholesterol, glucose, lipoprotein, PSA, testosterone levels and for responses to the Sexual Health Inventory for Men - SHIM, all part of usual care.
5. Research Method:

   We propose a prospective randomized control trial. Over twelve months, a sample of 100 English-speaking people, who are scheduled to start androgen deprivation therapy or have started within the last 7 days for prostate cancer at will be recruited for the study. Every two consented participants (and their partners if available) will be randomized. Therefore, one patient/partner will receive the intervention and one is placed in the control group. Both arms will receive the workbook and sexual counseling. The experimental group will also have access to an exercise and a nutrition program, with all three components supported by peer volunteers. Over the course of one month we predict eight patient/partners will be consented (four control, four intervention). Every four participants (and their partners if available) randomized to the intervention will form a group that will proceed through the program.

   Potential participants will be identified and invited by physicians. The Research Intern will consent participants. After consenting the participant will be instructed to bring their signed PAR-Q+ (24, 25) and consent form to the Introductory Meeting at the Prostate Centre. The research intern will also access participant's medical records to collect demographic information (cancer stage and treatment, co-morbidities, age) before they start the program.Participant's partners will also be invited to participate in the program The control group will attend the Introductory meeting and two sexual health counseling sessions .The intervention group will attend the Introductory meeting, the two sexual health meetings plus the exercise component (eight weekly exercise sessions) and the nutrition component (four monthly nutrition sessions) over a period of 6 months. A peer volunteer will be assigned to each intervention couple and will provide support during the intervention to help maintain participant's adherence to physical activity and healthy eating goals.Both intervention and control groups will provide measurements at each sexual health session (body-mass index -BMI, waist circumference, grip strength, blood pressure and heart rate) , describe their medical history and current medications. Both groups will attend follow-up measurement sessions at 12 and 24 months after baseline. Participants and their partners will fill out separate questionnaires at baseline, 6 months and at the two follow-up measurement sessions Participants and their partners will be interviewed at baseline, six, twelve, and twenty-four months. Interviews will be conducted until saturation at baseline (expected n=10) and the same couples will be interviewed again at the other time points. During these interviews qualitative data will be collected and transcribed for analysis. Questions related to their current physical activity experience, nutritional habits and barriers to maintaining a healthy diet and regular physical activity routine will be asked. In addition interviews with intervention participants will ask questions related to participants' satisfaction with the timing, quality, relevance & usefulness of topics discussed during the physical activity and nutrition sessions, motivation provided by instructors and peer volunteers and overall feedback about the program.
6. Statistical Analysis:

The Statistical Package for the Social Sciences (SPSS) version 14.0 (SPSS Inc., Chicago, IL) will be used for the statistical analysis. Significance will be set at P = 0.05 (two-tailed). Descriptive statistics [mean ± standard deviation (SD)] will be calculated for all characteristics. Differences between groups will be examined using Mann-Whitney U-test or Kruskal-Wallis test. A sample size calculation was based on the Quality of Life primary outcome measured by the FACT-P questionnaire (36). Change in quality of life will be determined by calculating change scores between different time-points. Considering mean score difference of 5, at the 5% level (2-tailed) and 80% power, a sample size of 41 should yield significant statistical differences. Based on our clinical and research experience with this population, we estimate recruiting about 50 patients per group in 12 months. Qualitative data will be systematically organized and sorted using ATLAS.ti 6.2 and analyzed through thematic analysis.

ELIGIBILITY:
Inclusion Criteria:

* All prostate cancer patients registered with BCCA-VIC or referred by an urologist that are prescribed to receive androgen deprivation in their care plan (not currently on hormone therapy)
* Must provide written, informed consent
* Must be able to understand, speak, read and write English, and have the cognitive capacity to complete written questionnaires
* Must be deemed ready to become more physically active, as determined by the PAR-Q+ and, if required, screened by a Canadian Society for Exercise Physiology Certified Exercise Physiologist® (CSEP-CEP) or medical doctor.
* Must be willing and able to attend the introductory meeting with the Prostate Centre nurse (baseline measurement recordings), 8 weeks of supervised exercise, 4 monthly nutrition meetings, two sexual health meetings (which includes measurement recording sessions at 6 months), and follow up at 12 and 24 months
* Must have access to a telephone
* Must be able to commit to the full 6 month intervention period of the study (i.e. no scheduled, extended absences) and follow up at 12 and 24 months. This does not preclude any participants from withdrawing from the study at any point.
* Must have greater than 12 months life expectancy

Exclusion Criteria:

* Prior invasive malignancy (except non-melanomatous skin cancer) or superficial bladder cancer unless disease free for a minimum of 5 years [for example, carcinoma in situ of the oral cavity is permissible]
* Previous hormone therapy within the past 5 years
* Participants who do not meet the following PAR-Q+(26, 27) criteria will be excluded from the study:
* Must not have a YES response to Q2 on pg1: Do you feel pain in your chest at rest, during your daily activities of living, OR when you do physical activity?
* Must not have a YES response to Q7 on pg 1: Has your doctor ever said that you should only do medically supervised physical activity?
* Must not have YES response to any sub-questions on pages 2-3 related to musculoskeletal conditions, diabetes, heart disease, mental health problems or learning difficulties, pulmonary conditions, spinal cord injury, stroke unless clearance is provided by a CSEP-CEP . A CSEP-CEP will only provide clearance to a positive response if upon further query it is determined that the participant is asymptomatic and the benefits of light to moderate intensity exercise outweigh any foreseeable health and injury risks. In such cases where the CSEP-CEP makes a professional determination that the foreseeable risks may outweigh the benefits of exercise or the participant does not know the necessary details of his or her own medical condition, then the participant will need to obtain clearance via the physician referral letter.
* PARQ+ form must be signed and dated within 6 months of entry into study
* More than 80 years of age

Max Age: 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in participant's quality of life on the Functional Assessment of Chronic Illnesses Therapy (FACT-P) | Baseline, 6 months, 12 months and 24 months
  Functional Assessment of Chronic Illnesses Therapy is a quality of life questionnaire for patients.with prostate cancer.
Change from baseline in patient's partner quality of life on the Quality of Life Scale (QOLS) | Baseline, 6 months,12 months, 24 months
  The Quality of Life Scale is a quality of life questionnaire that will be used for participants partners.
Change from baseline in fatigue on the Functional Assessment of Chronic Illnesses Therapy- Fatigue (FACIT-fatigue) | Baseline, 6 months, 12 months, 24 months
  The Functional Assessment of Chronic Illnesses Therapy is a measure of fatigue. This outcome will be tested for both participants and their partners.

SECONDARY OUTCOMES:
Change from baseline in intimacy on the Dyadic Adjustment Scale (DAS) | Baseline, 6 months, 12 months, 24 months
  The Dyadic Adjustment Scale is to measure intimacy. Both participants and their partners will complete this measure.

OTHER OUTCOMES:
Change from baseline in Body-Mass Index | Baseline, 3 months, 6 months, 12 months and 24 months
  Patient's weight and height will be measured at each meeting with the nurse. Body-Mass index [mass(kg)/height (m)2] will be calculated at each time point
Change from baseline in waist circumference | Baseline, 3 months, siz months, 12 months and 24 months
  Patient's waist circumference will be measured at each meeting with the nurse.
Change from baseline in grip strength | Baseline, 3 months, 6 months, 12 months and 24 months
  Patient's grip strength will be measured at each meeting with the nurse.
Changes from baseline in systolic blood pressure | Baseline, 3 months, 6 months, 12 months and 24 months
  Patient's blood pressure will be measured at each meeting with the nurse.
Change from baseline on blood levels of cholesterol, low density lipoprotein (LDL), high density lipoprotein (HDL), total glucose (TG), fasting glucose and glycated hemoglobin (HbA1) | Baseline, 12 and 24 months
  Blood measures will be obtained from patient's health records. Blood measures obtained within 12 months prior to starting the program will be used as baseline. Monitoring of these parameters are part of the standard of care.
Change in erectile dysfunction from baseline on the Sexual Health Inventory for Men (SHIM) | Baseline, 3 months, 6 months, 12 months and 24 months
  SHIM results will be obtained from patient's health records. Monitoring erectile dysfunction using this tool is part of the usual care.
Perceptions of patients and partners about the impact of the program on their psychosocial health assessed though qualitative interviews and program's meetings | Baseline, 6 months, 12 months, 24 months
  Interviews will be conducted until saturation at baseline (expected n=10) and the same couples will be interviewed again at the other time points. During these interviews qualitative data will be collected and transcribed for analysis. Questions related to their current physical activity experience, nutritional habits and barriers to maintaining a healthy diet and regular physical activity routine will be asked. In addition interviews with intervention participants will ask questions related to participants' satisfaction with the timing, quality, relevance & usefulness of topics discussed during the physical activity and nutrition sessions, motivation provided by instructors and peer volunteers and overall feedback about the program.
Operational impact of the program assessed though interviews with participants, peer-support volunteers, and health care providers and program documentation | Baseline, 3 months and 6 months
  • Operational impact - assessed though interviews with participants, peer-support volunteers, and health care providers, as well as any documentation related to the availability of space and personnel to conduct the program. Finally, direct costs of the program (ie. average salaries of qualified exercise professionals, materials, fitness equipment, etc.) will be obtained from available government economic data and project's expenditures.
Change from baseline on blood levels of Prostate-specific antigen (PSA) and testosterone | Baseline, 3 months, 6 months, 12 months, 24 months
  Blood measures will be obtained from patient's health records. Blood measures obtained within 12 months prior to starting the program will be used as baseline. Monitoring of these parameters are part of the standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Goulart, MD, Principal Investigator — British Columbia Cancer Agency; Satnam Sidhu, RD, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- BC Cancer Agency, Victoria, British Columbia, Canada